CLINICAL TRIAL: NCT00715286
Title: Neoadjuvant Chemotherapy (NACT) Followed by Interval Debulking Surgery vs Upfront Surgery Followed by Chemotherapy (CT) in Advanced Epithelial Ovarian Carcinoma (EOC): A Prospective Randomized Study
Brief Title: Neoadjuvant Chemotherapy in Advanced Epithelial Ovarian Cancer (EOC): A Phase III Randomized Study
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Prof Lalit Kumar, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I473
Record Dates: First submitted 2008-07-14; First posted 2008-07-15 (Estimated); Last update posted 2008-07-15 (Estimated); Status verified 2008-07

CONDITIONS: Ovarian Carcinoma
Keywords: epithelial ovarian cancer; neoadjuvant chemotherapy; randomized study
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Conventional arm: primary surgery followed by chemotherapy
  Interventions: Other: timing of surgery
- B (Experimental): Neoadjuvant chemotherapy followed by interval debulking
  Interventions: Other: timing of surgery

INTERVENTIONS:
Other: timing of surgery — Surgery is followed by chemotherapy
  Arms: A
Other: timing of surgery — Chemotherapy is followed by surgery
  Arms: B

SUMMARY:
To determine the impact of Neoadjuvant chemotherapy on surgical debulking rate, overall and disease-free survival and quality of life (QOL) in patients with advanced EOC.

ELIGIBILITY:
Inclusion Criteria:

* Age:20 to 65 years
* Epithelial ovarian carcinoma
* Stage IIIc & IV (pleural effusion only)
* ECOG PS 0-2
* Cytology/biopsy positive patients
* Good compliance
* Previously untreated patients

Exclusion Criteria:

* Any medical contraindication of surgery
* Psychiatric illness
* Cardiac, liver or renal dysfunction

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2001-11; Primary Completion 2007-04 (Estimated); Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
to compare the optimal debulking rate in primary surgery group and neoadjuvant chemotherapy group | post surgery

SECONDARY OUTCOMES:
post operative morbidity | 3 weeks post op

CONTACTS AND LOCATIONS:
Overall Officials: Lalit Kumar, DM, Principal Investigator — All India Institute of Medical Sciences
Locations (1):
- All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi, India